CLINICAL TRIAL: NCT02188953
Title: Evaluation of the Effectiveness, Acceptability, and Palatability of Air Classified Calcium Silicate (ACCS100) Clay to Reduce Aflatoxin Exposure in a High-risk Community in Kenya
Brief Title: Evaluation of ACCS100 to Reduce Aflatoxin Exposure in Kenya
Acronym: ACCS100
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kenya Medical Research Institute (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Texas A&M University (Other); Kenya Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Dr. John Vulule, Director, Center for Global Health Research, Kenya Medical Research Institute
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SSC Protocol No. 2603
Record Dates: First submitted 2014-07-02; First posted 2014-07-14 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Aflatoxicosis
Keywords: aflatoxin; Kenya
MeSH Terms: conditions — Aflatoxin Poisoning | interventions — ACCS100

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACCS100 (Experimental): Participants will consume 1 gram of ACCS100 at each meal (up to three times per day) for seven days. The ACCS100 will be administered by mixing a powder sachet into water.
  Interventions: Drug: ACCS100
- Calcium carbonate (Placebo Comparator): Participants will consume 1 gram of calcium carbonate at each meal (up to three times per day) for seven days. The calcium carbonate will be administered by mixing a powder sachet into water.
  Interventions: Drug: Calcium carbonate placebo

INTERVENTIONS:
Drug: ACCS100 — ACCS100 is made from Hydrated Sodium Calcium Aluminosilicate, which is a substance generally recognized as safe by the U.S. FDA.
  Other Names: Air Classified Calcium Silicate
  Arms: ACCS100
Drug: Calcium carbonate placebo
  Arms: Calcium carbonate

SUMMARY:
The purpose of this study is to pilot test the effectiveness, acceptability, and palatability of ACCS100 in a high-risk Kenyan population.

DETAILED DESCRIPTION:
Aflatoxins are harmful by-products of the molds Aspergillus flavus and A. parasiticus and are major contaminants of agricultural produce such as maize. Acute aflatoxin exposure (i.e., aflatoxicosis) can lead to jaundice, vomiting, abdominal pain, and liver failure, with documented fatality rates as high as 40%. Kenya experiences extreme aflatoxin exposure and fatal, recurring aflatoxicosis outbreaks. Numerous clinical trials have found heat processed calcium dioctahedral smectite clay [i.e., Air Classified Calcium Silicate (ACCS100)] to be safe and effective in binding to aflatoxin to decrease bioavailability and subsequently reduce toxin-induced effects. The investigators propose to pilot test the effectiveness, acceptability, and palatability of ACCS100 in a high-risk Kenyan population. If successful, ACCS100 could be scaled-up for use in Kenya to prevent aflatoxin-associated mortality during high-risk periods. To accomplish this objective, the investigators will recruit fifty health adults into a crossover study. Each participant will spend one week consuming ACCS100 and one week consuming a calcium carbonate placebo. Daily first morning void urine samples will monitor effectiveness in reducing aflatoxin bioavailability, and periodic questionnaires will assess acceptance and palatability.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years of age
* Consumes corn- and/or peanut-derived foods at least four times per week
* No plans to travel away from the household for more than one day in the next month

Exclusion Criteria:

* Women who may be pregnant
* History of medical illnesses
* Presence of protein or glucose in urine using chemstrip
* Does not provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline of urine aflatoxin M1 levels | Daily during each study arm
  Urine samples will be collected at baseline (Day 0) and daily for seven days during Arm 1 (Days 1-7). Urine samples will also be collected at baseline (Day 13) and daily for seven days during Arm 2 (Days 13-19).

SECONDARY OUTCOMES:
Serum aflatoxin B1-lysine adduct levels | Baseline of Arm 1 (Day 0) and end of arm 2 (Day 20)
  Baseline of Arm 1 (Day 0) and end of arm 2 (Day 20).
Palatability questionnaire | End of arm 1 (Day 8) and end of arm 2 (Day 20)
  End of arm 1 (Day 8) and end of arm 2 (Day 20)
Daily diary and adverse event reporting form | Daily during arm 1 (Days 2-8) and arm 2 (Days 14-20)
  Daily during arm 1 (Days 2-8) and arm 2 (Days 14-20)
Acceptability questionnaire | End of arm 2 (Day 20)
  End of arm 2 (Day 20)

CONTACTS AND LOCATIONS:
Overall Officials: John Vulule, PhD, Principal Investigator — Kenya Medical Research Institute; Ellen Yard, PhD, Principal Investigator — U.S. Centers for Disease Control and Prevention; Johnni Daniel, MPH, Principal Investigator — U.S. Centers for Disease Control and Prevention; Timothy Philips, PhD, Principal Investigator — Texas A&M University; Samuel Amwayi, MD, Principal Investigator — Kenya Ministry of Public Health and Sanitation
Locations (1):
- Makindu Health Center, Makindu, Kenya

REFERENCES:
- [Background] Wang P, Afriyie-Gyawu E, Tang Y, Johnson NM, Xu L, Tang L, Huebner HJ, Ankrah NA, Ofori-Adjei D, Ellis W, Jolly PE, Williams JH, Wang JS, Phillips TD. NovaSil clay intervention in Ghanaians at high risk for aflatoxicosis: II. Reduction in biomarkers of aflatoxin exposure in blood and urine. Food Addit Contam Part A Chem Anal Control Expo Risk Assess. 2008 May;25(5):622-34. doi: 10.1080/02652030701598694. PMID 18478481
- [Background] Phillips TD, Afriyie-Gyawu E, Williams J, Huebner H, Ankrah NA, Ofori-Adjei D, Jolly P, Johnson N, Taylor J, Marroquin-Cardona A, Xu L, Tang L, Wang JS. Reducing human exposure to aflatoxin through the use of clay: a review. Food Addit Contam Part A Chem Anal Control Expo Risk Assess. 2008 Feb;25(2):134-45. doi: 10.1080/02652030701567467. PMID 18286403
- [Background] Afriyie-Gyawu E, Wang Z, Ankrah NA, Xu L, Johnson NM, Tang L, Guan H, Huebner HJ, Jolly PE, Ellis WO, Taylor R, Brattin B, Ofori-Adjei D, Williams JH, Wang JS, Phillips TD. NovaSil clay does not affect the concentrations of vitamins A and E and nutrient minerals in serum samples from Ghanaians at high risk for aflatoxicosis. Food Addit Contam Part A Chem Anal Control Expo Risk Assess. 2008 Jul;25(7):872-84. doi: 10.1080/02652030701854758. PMID 18569006
- [Background] Wang JS, Luo H, Billam M, Wang Z, Guan H, Tang L, Goldston T, Afriyie-Gyawu E, Lovett C, Griswold J, Brattin B, Taylor RJ, Huebner HJ, Phillips TD. Short-term safety evaluation of processed calcium montmorillonite clay (NovaSil) in humans. Food Addit Contam. 2005 Mar;22(3):270-9. doi: 10.1080/02652030500111129. PMID 16019795
- [Background] Afriyie-Gyawu E, Mackie J, Dash B, Wiles M, Taylor J, Huebner H, Tang L, Guan H, Wang JS, Phillips T. Chronic toxicological evaluation of dietary NovaSil clay in Sprague-Dawley rats. Food Addit Contam. 2005 Mar;22(3):259-69. doi: 10.1080/02652030500110758. PMID 16019794
- See also: Description of ACCS100 clay — http://yourclay.com/